CLINICAL TRIAL: NCT06579976
Title: Multimodal High-frequency Ultrasound-based Study of Plaque Psoriasis Severity Index：a Prospective Cohort Study
Brief Title: Multimodal High-frequency Ultrasound-based Study of Plaque Psoriasis Severity Index
Status: Not yet recruiting | Type: Observational
Sponsor: Shanghai Yueyang Integrated Medicine Hospital (Other)
Responsible Party: Sponsor
Other Study IDs: 20230701
Record Dates: First submitted 2024-08-17; First posted 2024-08-30 (Actual); Last update posted 2024-08-30 (Actual); Status verified 2024-08

CONDITIONS: Plaque Psoriasis

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- psoriasis lesion area: Assessment of lesions in patients with plaque psoriasis using high-frequency ultrasound and local PASI scores
  Interventions: Other: No intervention
- non-psoriasis lesion area: Assessment of 2 cm next to lesions in patients with plaque psoriasis using high-frequency ultrasound
  Interventions: Other: No intervention

INTERVENTIONS:
Other: No intervention — This is an observational study, no intervention will be implemented.

SUMMARY:
Psoriasis (PsO) is a common chronic relapsing inflammatory disease, induced by a combination of genetic and environmental effects, which seriously affects the quality of life of patients.Psoriasis Area and Severity Index（PASI score ） ，as the most common method used by clinicians to assess the severity of psoriasis and the effectiveness of treatment, has the disadvantage of being subjective and superficial.We are therefore committed to establishing an objective, real-time, repeatable, non-invasive, microscopic assessment using high-frequency ultrasound. This study will use high-frequency ultrasound to detect the patient's lesion site and the 2cm site next to the lesion once, and the study will continue to recruit for 6 months.

DETAILED DESCRIPTION:
High-frequency ultrasound (HFUS) with a center frequency of more than 10 MHz, and a resolution of 16-158 μm. The detailed detection items are epidermal thickness (unit mm), dermal thickness (unit mm), hypoechoic cord thickness between epidermis and dermis (unit mm), epidermal echo intensity, dermal echo intensity, clarity of the boundary between dermis and subcutaneous tissue detected by Grayscale ultrasound; blood flow signal (pcs) detected by Color Doppler imaging and Power doppler imaging. The 8 tests will be detected the skin lesions and 2cm beside skin lesions area.Based on the correlation between the 8 indexes and local PASI scores, we will establish a model for the evaluation of psoriasis by multimodal high-frequency ultrasound.This study will use high-frequency ultrasound to detect the patient's lesion site and the 2cm site next to the lesion once, and the study will continue to recruit for 6 months

ELIGIBILITY:
Inclusion Criteria:

1. Patients who meet the medical criteria for plaque psoriasis
2. Those who voluntarily participate in this study and sign the informed consent form

Exclusion Criteria:

1. Patients with other types of psoriasis
2. Those with other active medical conditions that may affect assessment
3. During a severe uncontrollable acute or chronic local or systemic infection
4. Those with severe mental illness, cognitive impairment, and incapacity for personal behavior that makes them unsuitable to participate in a clinical study
5. Other reasons the investigator considers unsuitable for participation in this study

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients aged 18-75 years with plaque psoriasis who meet inclusion and exclusion criteria
Sampling Method: Non-Probability Sample
Enrollment: 45 (Estimated)
Dates: Start 2024-09-01 (Estimated); Primary Completion 2025-02-28 (Estimated); Study Completion 2025-05-01 (Estimated)

PRIMARY OUTCOMES:
High Frequency Ultrasound | Measurement of the patient's lesion and non-lesion areas were taken once 1 day
  epidermal thickness (unit mm) detected by Grayscale ultrasound
High Frequency Ultrasound | Measurement of the patient's lesion and non-lesion areas were taken once 1 day
  dermal thickness (unit mm) detected by Grayscale ultrasound
High Frequency Ultrasound | Measurement of the patient's lesion and non-lesion areas were taken once 1 day
  hypoechoic cord thickness between epidermis and dermis (unit mm) detected by Grayscale ultrasound
High Frequency Ultrasound | Measurement of the patient's lesion and non-lesion areas were taken once 1 day
  epidermal echo intensity detected by Grayscale ultrasound
High Frequency Ultrasound | Measurement of the patient's lesion and non-lesion areas were taken once 1 day
  dermal echo intensity detected by Grayscale ultrasound
High Frequency Ultrasound | Measurement of the patient's lesion and non-lesion areas were taken once 1 day
  clarity of the boundary between dermis and subcutaneous tissue detected by Grayscale ultrasound
High Frequency Ultrasound | Measurement of the patient's lesion and non-lesion areas were taken once 1 day
  blood flow signal (pcs) detected by Color Doppler imaging
High Frequency Ultrasound | Measurement of the patient's lesion and non-lesion areas were taken once 1 day
  blood flow signal (pcs) detected by Power doppler imaging

SECONDARY OUTCOMES:
Localized PASI | Measurement of the patient's lesion areas were taken once 1 day
  Same scoring criteria as PASI scores without area factors.

CONTACTS AND LOCATIONS:
Locations (1):
- Shanghai Yueyang Integrated Medicine Hospital, Shanghai, Shanghai Municipality, China

IPD SHARING:
Plan to Share IPD: No